CLINICAL TRIAL: NCT05812820
Title: Research of Change of Microbial System Intestines and Efficacy for Probiotic Treatment of Persistent Diarrhea in Children
Brief Title: Effects of Probiotic in Treatment of Persistent Diarrhea in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Children's Hospital, Vietnam (Other)
Responsible Party: Principal Investigator, Ha Dang Thuy, Deputy Head of Gastrointestinal Department, National Children's Hospital, Vietnam
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9720109
Record Dates: First submitted 2023-03-25; First posted 2023-04-14 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-07

CONDITIONS: Diarrhea
Keywords: Bacillus spore; Bacterial; Children; Gut microbiota; Persistent diarrhea; Viruses
MeSH Terms: conditions — Diarrhea; Virus Diseases

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: LiveSpo DIA30, LiveSpo CLAUSY, and RO water are indistinguishable in terms of smell. However, due to the opaque plastic container of the LiveSpo product suspension, the color and turbidity of the suspension are unrecognizable to investigators, except for the Principal Investigator (PI), analyzer, nurses, patient's parents, and patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Placebo Comparator): Control group receives the routine treatment and uses distilled water (RO) water
  Routine treatment at Department of Gastroenterology, Vietnam National Children's Hospital is as follows:
  * Antibiotics: oral (e.g. Zithromax® or Ciprofloxacin®) or intervention (ceftriaxone®, Ciprofloxacin®, Metronidazole®, Vancomycin®) drugs.
  * Oral rehydration Solution: Oremute
  * Zinc gluconate
  Interventions: Other: RO
- DIA30 (Experimental): DIA 30 group receives the routine treatment and uses distilled water plus B. subtilis, B. clausii and B. coagulans at 5 billion CFU/5 mL (LiveSpo® DIA 30)
  Routine treatment at Department of Gastroenterology, Vietnam National Children's Hospital is as follows:
  * Antibiotics: oral (e.g. Zithromax® or Ciprofloxacin®) or intervention (ceftriaxone®, Ciprofloxacin®, Metronidazole®, Vancomycin®) drugs.
  * Oral rehydration Solution: Oremute
  * Zinc gluconate
  Interventions: Combination Product: LiveSpo DIA30
- CLAUSY (Experimental): CLAUSY group receives the routine treatment and uses distilled water plus B. clausii at 2 billion CFU/5 mL (LiveSpo® CLAUSY)
  Routine treatment at Department of Gastroenterology, Vietnam National Children's Hospital is as follows:
  * Antibiotics: oral (e.g. Zithromax® or Ciprofloxacin®) or intervention (ceftriaxone®, Ciprofloxacin®, Metronidazole®, Vancomycin®) drugs.
  * Oral rehydration Solution: Oremute
  * Zinc gluconate
  Interventions: Combination Product: LiveSpo CLAUSY

INTERVENTIONS:
Combination Product: LiveSpo DIA30 — LiveSpo® DIA 30 has a registration number: 6547/2019/ĐKSP issued by the Food Safety Department of the Ministry of Health in Vietnam
  Arms: DIA30
Combination Product: LiveSpo CLAUSY — LiveSpo® CLAUSY has a registration number: 4071/2021/ĐKSP issued by the Food Safety Department of the Ministry of Health in Vietnam
  Arms: CLAUSY
Other: RO — Aquafina's distilled water and reverse osmosis (RO) water, produce by PepsiCo, have both obtained ISO 9001:2015 and ISO 22000:2018 certifications, which are internationally recognized standards for quality management and food safety management systems, respectively.
  The RO water ampoules are produced using a similar process as the LIVESPO DIA30/CLAUSY but contain 5ml of high-quality distilled water from Aquafina in an opaque plastic bottle
  Arms: Control

SUMMARY:
Persistent diarrhea is a common health problem worldwide, particularly in low-income countries. Approximately 3% to 20% of acute diarrhea episodes in children under 5 years of age become persistent diarrhea. Persistent diarrhea causes malnutrition, weight loss, and dehydration, as well as increasing treatment costs and the risk of mortality. One of the main causes of persistent diarrhea is the overgrowth and spread of bacteria, as well as viral infections that can disrupt the balance of microorganisms in the gut. Antibiotics are effective in treating bacterial infections that cause persistent diarrhea in children, but not against viral or parasitic infections. Overuse of antibiotics can lead to the growth of antibiotic-resistant bacteria, which poses a significant public health concern. Probiotics play a vital role in maintaining a healthy balance. Bacillus probiotic strains have an advantage over Lactobacillus probiotics as they can form spores that resist environmental stressors like heat, acid, and bile. This makes them more likely to survive the harsh conditions of the digestive tract and provide health benefits by reaching the intestines intact. Here, the investigators propose high-dose Bacillus spore probiotic supplementation as a potential solution for treating patients with persistent diarrhea.

The aim of the study is to assess the efficacy of two types of Bacillus probiotics which conclude LiveSpo CLAUSY (2 billion B. clausii) and LiveSpo DIA 30 (5 billion B. subtilis, B. clausii and B. coagulans) in supporting the treatment of children with persistent diarrhea.

Study Population: sample size is 150 patients and 30 healthy children. The study is carried out at Vietnam National Children's Hospital.

Description of Study Intervention: Totally 150 eligible patients are divided randomly into 3 groups (n = 50/group each): Patients in the Control group received the routine treatment and 2-3 times/day RO water while the patients in the probiotics group received 2-3 times/day LiveSpo DIA 30 or LiveSpo CLAUSY in addition to the same standard of care treatment. The standard treatment regimen is 5-9 days but can be extended further depending on the severity of the patient. Healthy children are grouped into the "Healthy" group solely for the purpose of comparing the microbiota between healthy children with those patients before and after treatment. Therefore, the Healthy group does not receive any intervention.

Study duration: 18 months

DETAILED DESCRIPTION:
Persistent diarrhea, which is defined as diarrhea that lasts for more than two weeks but less than four weeks, is a widespread health concern globally, particularly in low-income countries. It is a significant public health issue for children, especially in regions such as Asia, South America, and Africa. According to the World Health Organization (WHO), diarrhea is the second leading cause of morbidity and mortality in children after acute respiratory infections. Persistent diarrhea is a significant problem that defeats the nutritional status of children and increases treatment costs. The common pathogens associated with persistent diarrhea include:

Bacteria: Escherichia coli (E. coli), Campylobacter jejuni, Yersinia, Salmonella Enteritidis, Shigella spp., Clostridium difficile, Aeromonas.

Parasite: Giardia lamblia, Entamoeba histolytica, Cryptosporidium, Cyclospora, Microsporidia.

Viruses: norovirus, rotavirus, adenovirus. The intestinal microbiota serves as a protective barrier against pathogenic microorganisms and their toxins, playing a crucial role in the development and regulation of the immune system within the gut. Alterations in the gut microbiota have been observed in children with persistent diarrhea, highlighting its importance in maintaining gut health.

In terms of persistent diarrhea treatment, antibiotics are effective in treating bacterial infections that cause persistent diarrhea in children, but not against viral or parasitic infections. Overuse of antibiotics can lead to the growth of antibiotic-resistant bacteria, which poses a significant public health concern. Probiotics are live microorganisms that can provide health benefits to the host when consumed in sufficient amounts, playing a vital role in maintaining a healthy balance, which typically range from 1 to 10 billion per day, depending on the intended purpose of either prevention or supportive treatment. High-dose Lactobacillus rhamnosus GG probiotics, up to 40 billion per day, have been shown to be safe and effective in the treatment of antibiotic-associated diarrhea However, the quality of evidence is moderate to low. In comparison to Lactobacillus species, Bacillus species, such as B. subtilis, B. clausii, and B. coagulans, have the ability to form spores, which are resistant to environmental stressors such as heat, acid, and bile. This means that Bacillus probiotics are more likely to survive the harsh conditions of the digestive tract and reach the intestines intact, where they can provide health benefits. Bacillus probiotics have been found to be naturally resistant to certain antibiotics, which may make them a more effective option for individuals who are taking antibiotics or who have a history of antibiotic use. Thus, the investigators propose high-dose Bacillus spore probiotic supplementation as a potential solution for treating patients suffering from persistent diarrhea.

The overall aim of this study was to to assess the efficacy of two types of probiotics, the first one containing 2 billion B. clausii spores (LiveSpo® CLAUSY) per ampoule, and the second one containing 5 billion spores of three bacterial species per ampoule (LiveSpo® DIA 30), including Bacillus subtilis, B. clausii, and B. coagulans, in supporting the treatment of children with persistent diarrhea.

The first objective is evaluating the effectiveness of these products in alleviating typical symptoms and reducing the duration of treatment. The secondary objective is measuring changes in stool properties, major cytokine and IgA indices in stool and blood samples, and microbiota composition before and after treatment with LiveSpo® DIA 30 and LiveSpo® CLAUSY.

For this aim, the study is designed as a randomized, blind, and controlled clinical trial with 150 participants diagnosed with persistent diarrhea. The participants are randomized into 3 groups using permuted block randomization: a control group using RO water, experimental group 1 using LiveSpo® DIA 30 probiotics, and experimental group 2 using LiveSpo® CLAUSY probiotics. Each patient received 4-6 ampoules of the assigned probiotic product daily, divided into 2-3 doses after meals. The study included daily clinical assessment of indicators such as the number of types of stool, presence of mucus in stool, and frequency of daily bowel movements.

Contents and Methods for sub-clinical detection. The study participants were children aged 2 to 24 months who exhibited signs of loose stools or abnormal water on more than 3 occasions per day for a duration of between 14 and 30 days, diagnosed with persistent diarrhea, with no other systemic illnesses except diarrhea upon admission to the hospital and during treatment.

* Hematology and biochemical tests are conducted on day 0 only as part of routine procedures at the Hematology and Biochemistry Department of the National Children's Hospital.
* A multiplex Real-time RT PCR assay is conducted on day 0 only at the Department of Molecular Biology for Infectious Diseases of the National Children's Hospital to detect 24 intestinal pathogens in stool samples for the purpose of consulting on appropriate treatment therapy.
* A real-time PCR assay is conducted on stool samples on day 0 and 5 discharge day at the Spobiotic Research Center (proper noun) to detect probiotic spores, including B. subtilis, B. clausii, and B. coagulans, to cross-check the proper usage of probiotics or placebo in the experimental and control groups, respectively.
* ELISA tests are conducted on stool and blood samples on day 0 and 5 discharge day at the Department of Molecular Biology for Infectious Diseases of the Vietnam National Children's Hospital to determine proinflammatory cytokine levels and IgA and TNF-alpha levels, respectively, for evaluating changes in immune-related indicators during the treatment.
* The 16S V3-V4 metagenome sequencing analysis was carried out at Macrogen (Seoul, Korea) using next-generation sequencing (NGS) technology on the Illumina MiSeq platform (Illumina, San Diego, CA, USA), utilizing a 2 × 250 bp run configuration. DNA extracted from stool samples of about 5-10 representative patients from each group on day 0 and day 3 or/and day 7 was used for the analysis, with the goal of identifying changes in the microbiome.
* Data collection and statistical analysis involve the collection of individual medical records and the systematization of patient information into a dataset.

The investigators recommend that the CLAUSY and DIA30 groups continue using probiotics at the prevention dosage of 1-2 ampoules per day for an additional 28 days after discharge. Afterward, conduct a telephone interview with the parents of patients in all three groups (Control, CLAUSY, and DIA30) to inquire about any typical symptoms of diarrhea that may have recurred on Day 28 (optional).

The tabular analysis is performed on dichotomous variables using the χ2 test or Fisher's exact test when the expected value of any cell is below five. Continuous variables are compared using either the Wilcoxon test, t-test, or the Mann-Whitney test when data are not normally distributed. To determine if there was a statistically significant difference between three groups, an ANOVA test was performed. The correlations among the variables are assessed by Spearman's correlation analysis. Statistical and graphical analyses are performed on GraphPad Prism v8.4.3 software (GraphPad Software, CA, USA). The significance level of all analyzes is set at p < 0.05. P-values. The efficacy of LiveSpo® DIA 30 and LiveSpo® CLAUSY is evaluated and compared to the control based on the following clinical and sub-clinical criteria obtained from the Experiment and Control groups: Primary outcome: (i) Symptomatic relief duration diarrhea; Secondary outcomes: (ii) Regulate in the levels of cytokines such as IL-6, IL-8, IL-10, IL-17, IL-23 and TNF-alpha in blood samples. (iii) Decrease in the IgA level in blood and fecal samples. (iv) Improvement in the diversity and count of beneficial bacterial species compared to harmful bacteria species in the gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are between 2 months and 24 months old
* Have loose or unusual watery stools more than 3 times per day, lasting between 14 and 30 days
* Parents of the pediatric patient agree to participate in the study, explain and sign the research consent form

Exclusion Criteria:

* The patient had any systemic illness other than diarrhea on admission.
* Patient has any systemic complications during treatment.

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Changes in days of treatment for typical symptoms of persistent diarrhea | Day 0 to Day 12
  Changes in days of treatment for typical symptoms of persistent diarrhea, including:
  * the frequency of bowel movements per day (times/day)
  * the presence of mucus in stool (2 - lots of mucus, 1 - less mucus, 0 - no mucus)
  * the Bristol Stool Score ( 1 - Type 1, 2 - Type 2, 3 - Type 3, 4 - Type 4, 5 - Type 5A, 6 - Type 5B)

SECONDARY OUTCOMES:
Changes in presence of white blood cells and red blood cells by stool microscopy | Day 3 and Day 5 compared to Day 0
  Changes in presence of white blood cells (yes/no) and red blood cells (yes/no).
Changes in Intestinal microbiota | Day 3 or/and Day 7 compared to Day 0
  Changes in intestinal microbiota (bacterial species composition) in the stool samples of patients with persistent diarrhea before (Day 0) and after treatment (Day 3 or/and 7), as well as with that of healthy children (Day 0, no intervention)
Changes in cytokines levels of blood samples | Day 5 compared to Day 0
  Changes in levels (pg/mL) in several cytokines, including tumor necrosis factor-α (TNF-α), interleukin-6 (IL-6), interleukin-8 (IL-8), interleukin-10 (IL-10), interleukin-17 (IL-17), interleukin-23 (IL-23)
Changes in IgA levels in both stool and blood samples | Day 5 compared to Day 0
  Changes in levels (µg/mL) of pro-inflammatory IgA in both stool and blood samples
Change the stool pH values | Day 3 and Day 5 compared to Day 0
  Change the pH values of stool samples at day 3-5 (after treatment) compared with day 0 (before treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Dang T Ha, MD, Principal Investigator — Department of Gastroenterology, Vietnam National Children's Hospital
Locations (1):
- Department of Gastroenterology, Vietnam National Children's Hospital, Hanoi, Vietnam, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data or samples share that will be coded, with no PHI include. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a study protocol, informed consent form (ICF), clinical study report (CSR). For more information or to submit a request, please contact clinicaltrial.probiotics@gmail.com

REFERENCES:
- [Background] Sarker SA, Ahmed T, Brussow H. Persistent diarrhea: a persistent infection with enteropathogens or a gut commensal dysbiosis? Environ Microbiol. 2017 Oct;19(10):3789-3801. doi: 10.1111/1462-2920.13873. Epub 2017 Sep 14. PMID 28752952
- [Background] Fan Q, Yi M, Liu H, Wang Y, Li X, Yuan J, Wang L, Hou B, Li M. The Impact of Age and Pathogens Type on the Gut Microbiota in Infants with Diarrhea in Dalian, China. Can J Infect Dis Med Microbiol. 2020 Nov 30;2020:8837156. doi: 10.1155/2020/8837156. eCollection 2020. PMID 33312314
- [Background] Bandsma RHJ, Sadiq K, Bhutta ZA. Persistent diarrhoea: current knowledge and novel concepts. Paediatr Int Child Health. 2019 Feb;39(1):41-47. doi: 10.1080/20469047.2018.1504412. Epub 2018 Aug 6. PMID 30079818
- [Background] Szajewska H, Kolodziej M. Systematic review with meta-analysis: Lactobacillus rhamnosus GG in the prevention of antibiotic-associated diarrhoea in children and adults. Aliment Pharmacol Ther. 2015 Nov;42(10):1149-57. doi: 10.1111/apt.13404. Epub 2015 Sep 13. PMID 26365389
- [Background] Belkaid Y, Hand TW. Role of the microbiota in immunity and inflammation. Cell. 2014 Mar 27;157(1):121-41. doi: 10.1016/j.cell.2014.03.011. PMID 24679531
- [Background] Hill C, Guarner F, Reid G, Gibson GR, Merenstein DJ, Pot B, Morelli L, Canani RB, Flint HJ, Salminen S, Calder PC, Sanders ME. Expert consensus document. The International Scientific Association for Probiotics and Prebiotics consensus statement on the scope and appropriate use of the term probiotic. Nat Rev Gastroenterol Hepatol. 2014 Aug;11(8):506-14. doi: 10.1038/nrgastro.2014.66. Epub 2014 Jun 10. PMID 24912386
- [Background] Ugboko HU, Nwinyi OC, Oranusi SU, Oyewale JO. Childhood diarrhoeal diseases in developing countries. Heliyon. 2020 Apr 13;6(4):e03690. doi: 10.1016/j.heliyon.2020.e03690. eCollection 2020 Apr. PMID 32322707
- [Background] Abba K, Sinfield R, Hart CA, Garner P. Pathogens associated with persistent diarrhoea in children in low and middle income countries: systematic review. BMC Infect Dis. 2009 Jun 10;9:88. doi: 10.1186/1471-2334-9-88. PMID 19515227
- [Background] Olvera-Rosales LB, Cruz-Guerrero AE, Ramirez-Moreno E, Quintero-Lira A, Contreras-Lopez E, Jaimez-Ordaz J, Castaneda-Ovando A, Anorve-Morga J, Calderon-Ramos ZG, Arias-Rico J, Gonzalez-Olivares LG. Impact of the Gut Microbiota Balance on the Health-Disease Relationship: The Importance of Consuming Probiotics and Prebiotics. Foods. 2021 Jun 2;10(6):1261. doi: 10.3390/foods10061261. PMID 34199351
- [Background] Guo Q, Goldenberg JZ, Humphrey C, El Dib R, Johnston BC. Probiotics for the prevention of pediatric antibiotic-associated diarrhea. Cochrane Database Syst Rev. 2019 Apr 30;4(4):CD004827. doi: 10.1002/14651858.CD004827.pub5. PMID 31039287
- [Background] Tridip K. Das, Shrabani Pradhan, Sudipta Chakrabarti, Keshab Chandra Mondal, Kuntal Ghosh, Current status of probiotic and related health benefits, Applied Food Research, Volume 2, Issue 2, 2022, 100185, ISSN 2772-5022
- [Derived] Dang HT, Phung TTB, Tran DM, Bui ATP, Vu YH, Luong MT, Nguyen HM, Trinh HT, Vo HTN, Nguyen TTT, Nguyen AH, Tung PD, Tran LH, Van Nguyen AT. High-dose multi-strain Bacillus probiotics enhance treatment and reduce antibiotic usage in children with persistent diarrhea through immune and microbiota modulation. Sci Rep. 2025 Aug 18;15(1):30231. doi: 10.1038/s41598-025-15199-y. PMID 40826150
- [Derived] Dang HT, Tran DM, Phung TTB, Bui ATP, Vu YH, Luong MT, Nguyen HM, Trinh HT, Nguyen TT, Nguyen AH, Van Nguyen AT. Promising clinical and immunological efficacy of Bacillus clausii spore probiotics for supportive treatment of persistent diarrhea in children. Sci Rep. 2024 Mar 18;14(1):6422. doi: 10.1038/s41598-024-56627-9. PMID 38494525
- See also: Diarrheal disease — https://www.who.int/news-room/fact-sheets/detail/diarrhoeal-disease